CLINICAL TRIAL: NCT04906239
Title: The Effect of Bilateral Erector Spina Block on Postoperative Pain in Adult Cardiac Surgery: A Randomized, Clinical Study.
Brief Title: The Effect of Bilateral Erector Spina Plane Block on Postoperative Pain in Adult Cardiac Surgery.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kahramanmaras Sutcu Imam University (Other)
Responsible Party: Principal Investigator, Yavuz Orak, Assistant Professor, Kahramanmaras Sutcu Imam University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2020/18-10
Record Dates: First submitted 2021-05-17; First posted 2021-05-28 (Actual); Last update posted 2022-04-19 (Actual); Status verified 2022-04

CONDITIONS: Postoperative Pain; Opioid Use
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group ESP (Active Comparator): While the patient is in a sitting position, A ultrasound probe covered with a sterile sheath will be placed approximately 2 cm to the right or left of the T 4-5 spinous process. After the T 4-5 transverse process and the erector spinae muscle above it are shown, a quincke-type needle will be inserted into the skin at an angle of approximately 30 degrees from cranial to caudal with the entrance made using the in-plane technique. When the transverse process is touched, the needle will be pulled out and a local anesthetic solution will be applied to the fascia beneath the erector spinae muscle. A 20 mL dose of 0.25% bupivacaine, which has been shown to spread both above and below the T 4-5 level, will be injected.The same procedure will be repeated on the contralateral side of the T5 spinous process and half of the remaining bupivacaine dose will be injected. The total volume of bupivacaine injected on both sides will be 20 mL.
  Interventions: Procedure: Erector Spinae Plane Block
- Group Control (No Intervention): No block will be made to the control group.
  After extubation, 1mg / kg tramadol will be applied routinely to both groups, and PCA (Patient Control Analgesia) and morphine consumption and VAS (visual analog scale) pain scores of both groups will be evaluated and recorded at the 1st, 4th, 12th and 24th hour. When VAS is 3, patients will be advised to press the PCA device.

INTERVENTIONS:
Procedure: Erector Spinae Plane Block — A high-frequency ultrasound linear probe, covered with a sterile sheath, will be placed approximately 2 cm to the right or left of the T 4-5 spinous process. After showing the T 4-5 transverse process and the erector spinae muscle on top of it, a 22-gauge, 80 mm insulated quincke type needle will be inserted into the skin at an angle of approximately 30 degrees from cranial to caudal, using the in-plane technique. When the transverse process is touched, the needle will be pulled out and after a negative aspiration test with 0.5 mL of normal saline and after the demonstration of a hypo-echogenic image and hydro dissection, a local anesthetic solution will be applied to the fascia beneath the erector spinae muscle. A 20 mL dose of 0.25% bupivacaine, which has been shown to spread both above and below the T 4-5 level, will be injected.
  Arms: Group ESP

SUMMARY:
Failure to adequately prevent pain after heart surgery increases morbidity and results in a high incidence of persistent poststernotomy pain syndrome. Aim in this study is to investigate analgesic consumption and postoperative pain effect in patients who underwent cardiopulmonary bypass with Erector Spinae Block, a new block.

DETAILED DESCRIPTION:
Failure to adequately prevent pain after heart surgery increases morbidity and results in a high incidence of persistent poststernotomy pain syndrome.

The use of special opioid-based analgesia causes adverse effects such as nausea, vomiting, sedation, urinary retention, respiratory depression and delayed tracheal extubation.

Regional anesthesia techniques such as pectoralis nerve block and serratus anterior block provide analgesia in the sternum and protection from pain in the lateral / posterior chest wall.

Ketamine and a2 agonists were used for intravenous analgesia to reduce opioid consumption. However, these drugs have potential side effects that limit their extensive clinical use as analgesic agents. The use of regional anesthetic techniques, e.g. thoracic epidural and thoracic paravertebral block, dural puncture, epidural hematoma, spinal cord injury, hypotension, pneumothorax, epidural abscess, ipsilateral Horner's syndrome Their use has declined due to the high failure rate of as much as 15% (especially for the thoracic epidural) and the significant possibility of complications.

Erector spinae (ESP) block, a new method, provides a wide multi dermatomal sensory block. In the T 4-5 spinous process, the bilateral ESP block provides analgesia from T2 to T9 sensory level and results in both somatic and visceral analgesia by blocking both the dorsal and ventral of the spinal nerves, including the sympathetic chain. This block can provide sufficient analgesia for the median sternotomy because the main nerve supply to the sternal region is from T2 to T6. Our aim in this study is to investigate analgesic consumption and postoperative pain effect in patients who underwent cardiopulmonary bypass with Erector Spina Block, a new block.

ELIGIBILITY:
Inclusion Criteria:

* Male and / or female patients aged 18-65 will be included in the study.
* Normal left ventricular function (alternating one, two and three vessels).
* coronary artery patients scheduled for elective coronary artery surgery under cardiopulmonary bypass,
* Valvular diseases planned for elective valve replacement with normal left ventricular function, ASD (Atrial Septal Defect) cases for atrial septal defect closure, and patients without left ventricular dysfunction (E / F≥ 50-55%) elective valve + CABG will be included in the study.

Exclusion Criteria:

* Patients requiring acute coronary syndrome and emergency cardiovascular surgery,
* Patients who have had myocardial infarction within the past month
* Recurrent cardiovascular surgery
* Off-pump coronary artery bypass surgery (OPCAB)
* Patients with chronic inflammatory disease (rheumatoid arthritis, malignancy, psoriasis, etc.), autoimmune disease, immunocompromised patients
* Patients with chronic renal failure, liver disease, active infection
* Patients older than 80 years and smaller than 18 years
* Patients with coagulation disorders

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-02-15 (Actual); Study Completion 2022-03-15 (Actual)

PRIMARY OUTCOMES:
Morphine consumption by PCA (Patient Control Analgesia) | The change from baseline in the postoperative period 1, 4, 12 and 24 hours after extübation
  Morphine consumption used in case of pain

SECONDARY OUTCOMES:
Pain (VAS Score) | Change From Baseline of VAS Score at 1, 4, 12 and 24 hours after being extubated will be recorded.
  Change from Baseline VAS Score. from 1 to 10 , 0: No pain, 10: 10 pain that can not be tolerated

CONTACTS AND LOCATIONS:
Overall Officials: Yavuz Orak, MD, PhD, Principal Investigator — Kahramanmaraş Sütçü İmam Üniversitesi Tıp Fakültesi, Anesteziyoloji ve Reanimasyon Bölümü
Locations (2):
- Turkey (Türkiye) (2):
  - Kahramanmaras Sutcu Imam University Faculty of Medicine, Kahramanmaraş
  - Yavuz Orak, Kahramanmaraş

IPD SHARING:
Plan to Share IPD: No